CLINICAL TRIAL: NCT06272578
Title: A Cross-sectional Observational Cohort Study to Evaluate the Prevalence of Asymptomatic Cardiac Structural Abnormalities and Cardiac Dysfunction in a Contemporary Outpatient at Risk Population With Chronic Kidney Disease
Brief Title: Screen CardRen - A Cross-sectional Observational Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Univ.-Prof. Dr. med. Frank Edelmann, Prof. Dr. med. Frank Edelmann, Charite University, Berlin, Germany
Other Study IDs: 20021405
Record Dates: First submitted 2023-12-05; First posted 2024-02-22 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure; Chronic Kidney Diseases
MeSH Terms: conditions — Heart Failure; Renal Insufficiency, Chronic | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Fasting blood samples will be collected preferably from a cubital vein or any other vein of the upper extremity, if cubital veins are not accessible. The collected blood volume will comprise 12 ml for local baseline laboratory and another 12 ml for processing and storage for proteomic analyses.
  Biomaterial will be collected at single study visit for all participants and stored as frozen samples (-80°C) at the central biobanking facility (Zebanc) of Charité Campus Virchow Klinikum after immediate processing. Proteome measurement and analysis will be performed only after study enrolment has been closed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Echocardiography — Echocardiography

SUMMARY:
In this single-centre, cross-sectional study, the investigators aim to assess the prevalence of asymptomatic echocardiographic structural and functional cardiac abnormalities in adult CKD patients with additional cardiovascular risk factors. Furthermore, with the use of Olink technology, analyses of the plasma proteome will be performed to identify potential protein pathways associated with early structural changes.The investigators hypothesize that protein expression will be altered in patients with prevalent echocardiographic abnormalities that indicate stage B heart failure.

DETAILED DESCRIPTION:
Background/Rationale:

Chronic kidney disease and cardiovascular disease share a large set of risk factors, such as arterial hypertension, type 2 diabetes mellitus and dyslipidaemia. Chronic kidney disease, even in early stages, further increases the risk for cardiovascular diseases such as heart failure.

Objectives and Hypotheses:

In this single-centre, cross-sectional study, the investigators will aim to assess the prevalence of asymptomatic echocardiographic structural and functional cardiac abnormalities in adult CKD patients with additional cardiovascular risk factors. Furthermore, with the use of Olink technology, analyses of the plasma proteome will be performed to identify potential protein pathways associated with early structural changes. The investigators hypothesize that protein expression will be altered in patients with prevalent echocardiographic abnormalities that indicate stage B heart failure.

Methods:

Study design: single-centre, cross-sectional, non-interventional study Data Source(s): electronic case report form containing patient history, clinical status and physical examination, imaging data from echocardiography, air displacement plethysmography data, plasma proteome data obtained from Olink technology-based analysis of blood samples Study Population: Adult chronic kidney disease patients with additional cardiovascular risk factors (at least one of the following: arterial hypertension, type 2 diabetes mellitus, and dyslipidaemia). The inclusion criteria are further defined in the corresponding section of the study protocol.

Exposure(s): chronic kidney disease and cardiovascular risk factors such as arterial hypertension, type 2 diabetes mellitus, dyslipidaemia, or atherosclerotic vascular disease

Outcome(s):

Primary objective:

• Assess the frequency of stage B heart failure as indicated by structural or functional cardiac abnormalities assessed by echocardiography and/or corresponding laboratory parameters

Secondary objectives:

* Identification of possible predictive parameters for significant cardiac dysfunction (Heart Failure Stage B) in a contemporary at risk cohort with renal dysfunction, based on imaging and proteomics data
* Building of the Berlin-Brandenburg prevention network to improve the intersectional cooperation to identify, diagnose and follow-up risk patients
* Establishment of tools like US.2 AI, electronic health records, central data management in order to enable a fast construction while working resource-friendly
* Follow-up of risk patients based on mobile sensors/apps
* Adoption of screening in standard care Sample Size Estimations: The study is focused on the estimation of the prevalence of significant asymptomatic cardiac structural abnormalities and cardiac dysfunction in a contemporary at risk cohort with chronic kidney disease. Therefore, the investigators will calculate the corresponding two-sided 95% confidence interval. With a sample size of 400 patients, a two-sided 95% confidence interval for an assumed prevalence of 30% can be determined with an extension of ± 4%.

Statistical Analysis:

Objectives will be analyzed according to their scaling and distribution characteristics, including appropriate descriptive location and variability parameters and 95% confidence intervals. Additionally, multiple regression analyses will be performed in order to identify potential risk factors for significant cardiac dysfunction.

ELIGIBILITY:
Inclusion Criteria:

Chronic Kidney Disease, stages G1-G4, AND

* Estimated glomerular filtration rate (eGFR) as determined by the 2009 CKD-EPI Cr equation ≥ 60 ml/min/1.73m², if UACR ≥30 mg/g (≥3 mg/mmol) OR
* eGFR according to CKD-EPI 2009 Cr equation < 60 ml/min/1.73m², but > 15 ml/min/1.73m²

Diabetes mellitus type 2 OR

* Pathological findings in oral glucose tolerance test (≥ 200 mg/dl (2h)) OR
* documented HbA1c ≥ 6.5 % OR
* Intake of any antidiabetic medication (in case of previously established diagnosis of Diabetes mellitus type 2) OR
* Fasting blood glucose ≥ 126 mg/dl

Arterial Hypertension Grade ≥ 1 OR

* Blood pressure of ≥ 140/90 mmHg, defined according to the 2018 ESC guidelines on arterial hypertension (Williams) OR
* Intake of antihypertensive drugs

Hypercholesterolemia OR

* LDL-cholesterol > 130mg/dl OR
* Intake of a lipid-lowering medication initiated to treat dyslipoptroteinemia

Exclusion Criteria:

History of acute kidney injury > stage 1 according to KDIGO criteria in the two weeks prior to study visit

* Chronic kidney disease Stage 5 (end-stage renal disease)
* Previous diagnosis of chronic heart failure
* Acute myocardial infarction in the past 30 days prior to study visit
* Stroke in the past 30 days prior to study visit
* Known congenital heart disease
* Previous diagnosis of a specific cardiomyopathy, infiltrative cardiac disease, pericardial constriction, sarcoidosis, amyloidosis and other storage diseases
* Implanted cardiac devices, such as pacemakers, implantable cardioverter-defibrillators, cardiac resynchronization devices
* Implanted mechanical valve prosthesis
* Inability to give informed consent
* Lack of health insurance
* Organ transplanted
* Intake of immunosuppressive medication
* Major surgery in the 6 months before study visit, such as cardiac bypass surgery or valve replacement surgery (thoracotomy), major vascular surgery (such as replacement of aortic root, ascending part, aortic arch or any part of the abdominal aorta), major abdominal surgery (e.g. Whipple procedure, colorectal resection, gastrectomy and others) or limb amputation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise 400 adult patients with chronic kidney disease, defined as elevated urine albumin to creatinine ratio (UACR > 30 mg/g or >3 mg/mmol) or reduced estimated glomerular filtration rate (eGFR < 60 ml/min/1.73m²) at a one-time measurement.
  In addition to renal function impairment, study participants will either have a background of cardiovascular risk factors, including arterial hypertension, type 2 diabetes mellitus or hypercholesterolemia.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-02-27 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
prevalence of significant asymptomatic cardiac structural abnormalities and cardiac dysfunction | 1 year
  Transthoracic echocardiographic measurements are the primary outcome parameters and will be conducted according to the current recommendations for cardiac chamber quantification of the American Society of Echocardiography and the European Association of Cardiovascular Imaging, the latest update on left ventricular diastolic function assessment and recommendations on aortic stenosis quantification.
Proteomic analysis | 1 year
  Proteomic analysis will be performed using Olink technology, which is based on proximity extension assay (PEA) technology combined with next generation sequencing. This method has demonstrated accuracy and sensitivity in detecting minute quantities of proteins (sub-pg/ml), making it suitable for conducting extensive multiplex assays covering a wide dynamic range. In this study, plasma samples

SECONDARY OUTCOMES:
Duration of echocardiographic examination | 1 year
  The duration of echocardiographic examination as mean, median, standard deviation, quantiles and range in comparison between portable and cart-based device
Time saved by portable echocardiography and automated image analysis | 1 year
  Amount of time savings in minutes as mean, median, standard deviation, quantiles and range in comparison between portable device and automated image analysis, potential impact on waiting period for patients requiring echocardiography
Image quality of cart-based vs. portable echo images | 1 year
  The number of echocardiographic examinations with acceptable image quality as frequencies and percentages in comparison between devices

CONTACTS AND LOCATIONS:
Overall Officials: Frank Edelmann, Prof. Dr., Principal Investigator — German Heart Institute
Locations (1):
- German Heart Center Charité (DHZC), Wedding, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No